CLINICAL TRIAL: NCT04868045
Title: Evaluation of The Development of Central Resistance to Thyroid Hormone After Prolonged Exposure to Excess Thyroid Hormone in Thyroid Cancer Patients
Brief Title: Study of Resistance to Thyroid Hormone After Long-term Exposure in People With Thyroid Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-079
Record Dates: First submitted 2021-04-28; First posted 2021-04-30 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Thyroid Cancer
Keywords: Thyrotropin Releasing Hormone (TRH); 20-079
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Thyrotropin-Releasing Hormone; Thyroxine

STUDY DESIGN:
Intervention Model Description: This is a prospective, single center, pilot study of the hypothalamic-pituitary-thyroid axis in adult patients with thyroid cancer.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Patients with a history of thyroid hormone suppression (TSH<0.5 mU/L) for at least 5 years (Experimental): Study subjects will be given 200mcg of TRH as a single intravenous (IV) bolus in endocrine clinic on Day 1 and Day 5. LT3 will be administered orally, twice a day (12 hours apart i.e. 8 AM and 8 PM) at a dosage of 10 mcg on Day 2-4. Levothyroxine will be taken after the TRH stimulation tests on Day 1 and day 5. Levothyroxine will be taken on Days 2-4 of the study. *Patients will take their own LT4 that they are prescribed by their endocrinologist. The dose of Levothyroxine is titrated for each patient.
  Interventions: Drug: Thyrotropin Releasing Hormone (TRH); Drug: levothyroxine; Other: Hypothyroidism QOL questionnaire
- Patients with no history of TSH suppression (Experimental): Study subjects will be given 200mcg of TRH as a single intravenous (IV) bolus in endocrine clinic on Day 1 and Day 5. LT3 will be administered orally, twice a day (12 hours apart i.e. 8 AM and 8 PM) at a dosage of 10 mcg on Day 2-4. Levothyroxine will be taken after the TRH stimulation tests on Day 1 and day 5. Levothyroxine will be taken on Days 2-4 of the study. *Patients will take their own LT4 that they are prescribed by their endocrinologist. The dose of Levothyroxine is titrated for each patient.
  Interventions: Drug: Thyrotropin Releasing Hormone (TRH); Drug: levothyroxine; Other: Hypothyroidism QOL questionnaire

INTERVENTIONS:
Drug: Thyrotropin Releasing Hormone (TRH) — TRH administration will be given as a 200-mcg single IV bolus on Day 1 and Day 5.
Drug: levothyroxine — Patients maintenance dose of levothyroxine will be taken throughout the study. On Day
  1 and Day 5, the levothyroxine will be taken after the TRH test is complete. On Days 2- 4, the levothyroxine will be taken in the morning.
Other: Hypothyroidism QOL questionnaire — Administer standardized Hypothyroidism QOL questionnaire.

SUMMARY:
The purpose of this study is to find out whether people who have had thyroid cancer develop resistance to treatment with thyroid hormones after having received high doses of thyroid drugs for many years.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Due to a diagnosis of thyroid cancer, patient underwent a total thyroidectomy based on pathology.
* No evidence of active disease based on routine surveillance testing showing no suspicious findings on neck ultrasound and low thyroglobulin levels (≤1.0 ng/ml) with negative thyroglobulin antibodies within one year of study enrollment. For the study patients, this response can be evaluated after five years of TSH suppression. For control subjects, this response can be evaluated after two years of surveillance.
* Two groups:

  * 8 patients with a history of thyroid hormone suppression (TSH<0.5 mU/L) for at least 5 years
  * 8 patients with no history of TSH suppression
* Normal TSH level based on the laboratory reference range for at least 6 months at the time of study enrollment.
* Blood pressure range of >90/60 and <180/100. Patients may be included in the study if blood pressure has been treated with medication and normalized.

Exclusion Criteria:

* Patient reported history of symptomatic heart disease including unstable angina or NYHA stage III or IV heart failure.
* Patient reported history of one of the following cardiac arrhythmias: atrial fibrillation, atrial flutter, paroxysmal supraventricular tachycardia, ventricular fibrillation, or ventricular tachycardia.
* Patient reported history of uncontrolled hypotension (<90/60) or hypertension (>180/100).
* History of renal dysfunction with creatinine more than 1.5 times the upper limit of normal based on recent laboratory testing
* Known hypersensitivity to the drug
* Pregnant or breast feeding
* Prior history of seizures or brain damage
* Patients on chronic therapy with levodopa
* Patients on therapeutic doses of acetylsalicylic acid (2 - 3.6 gm/day)
* Patients with conditions that result in disruption of the hypothalamic-pituitary axis (i.e. hypophysectomy, hypopituitarism, pituitary tumor/surgery, head irradiation, or head trauma).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
change in peak TSH levels | day 5
  in response to TRH stimulation between day 1 (baseline) and day 5 after three days of high dose LT3 treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Fish, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm